CLINICAL TRIAL: NCT03908996
Title: Preliminary Trial to Evaluate the Effectiveness of the Profile by Sanford Weight Management Program in Endometrial Cancer Patients
Brief Title: the Effectiveness of a Weight Management Program in Patients Who Have Completed Treatment for Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH Profile II
Record Dates: First submitted 2018-08-14; First posted 2019-04-09 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Endometrial Cancer; Overweight
MeSH Terms: conditions — Endometrial Neoplasms; Overweight

STUDY DESIGN:
Intervention Model Description: All enrolled patients will participate in the Profile weight management program
Masking Description: A participant will not be informed of the analysis done on their stool samples. The results of the testing done on a participants stool sample will not be entered into the participants medical record.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Profile by Sanford (Experimental): All enrolled subjects are assigned to participate in the Profile by Sanford weight management program for a period of 12 months..Subjects will follow the Profile program and will be provided a nutritional plan which includes consuming Profile nutritional supplements and other food items. Subjects will work with a Profile lifestyle coach to develop a personalized nutrition plan, discuss their activity, and lifestyle behavior. Subjects on this research study will follow the Profile by Sanford weight loss and management plan as all Profile members. All enrolled subjects will collect and return a fecal specimen prior to beginning the Profile by Sanford weight management plan and again after 6 months of participation.
  Interventions: Behavioral: Profile by Sanford weight management plan

INTERVENTIONS:
Behavioral: Profile by Sanford weight management plan — The purpose of this study is to observe weight changes in patients who completed endometrial cancer treatment, are clinically overweight, and who participate in the Profile by Sanford weight management program. An exploratory purpose is to examine the bacterial content of the patient's gut by examining stool specimens before starting the Profile by Sanford weight management program and after 6 months of participation in the Profile by Sanford weight management program.

SUMMARY:
The primary purpose of this study is to evaluate the effectiveness of a 12-month comprehensive weight management program on weight change in overweight/obese patients following treatment for endometrial cancer. During the study period, subjects will be monitored for recurrence during routine clinic visits A secondary exploratory purpose of this study will be to evaluate the gut microbiome in this intervention group and the changes that may occur while participating in a weight loss and weight management program.

DETAILED DESCRIPTION:
All enrolled subjects will participate in the Profile weight loss and weight management program for a period of 12 months. They will work with a Profile lifestyle coach weekly to develop a personalized nutrition plan, discuss their activity, and lifestyle behavior as done with all Profile members. A comparison of similar retrospective chart reviews based on age, weight in pounds and stage of cancer will be conducted using the Electronic Medical Record (EMR). All enrolled subjects will collect and return a fecal specimen prior to beginning the weight management plan and again after 6 months of participation. The stool sample will be used to understand gut health.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older with a diagnosis of endometrial cancer
* No known metastatic disease
* Has completed all treatment for their endometrial cancer at least 2 months prior to enrollment.
* Has a BMI (Body Mass Index) of 30 or higher
* Ability to understand the purpose of study and willingness to sign consent
* Willingness to collect fecal specimens at the required time points
* Capable of following the dietary guidelines and instructions for the Profile weight management plan
* Agrees to sharing information between Profile and Sanford Research study personnel

Exclusion Criteria:

* BMI (Body Mass Index) less than 30
* Known metastatic disease
* Receiving treatment or expected to receive treatment for endometrial cancer or any other cancer
* Any psychological, familial, sociological conditions that the physician feels will interfere with medical follow-up and compliance on the study
* Taking insulin for diabetes (oral medications for diabetes allowed)
* Use of corticosteroids for a chronic medical condition
* Known liver disease
* Bowel or stomach disorders that the physician feels would interfere with Profile participation.
* Any history of malabsorption syndrome or substantial amounts of small bowel or stomach surgery that impairs nutrient absorption

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients who has a diagnosis of endometrial cancer and have completed standard of care treatment.
Enrollment: 25 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Determine weight change from baseline to 6 months. | 6 months after starting weight management program
  All enrolled subjects will be weighed in pounds and the difference from baseline to 6 months will be recorded.
Determine weight change from baseline to 12 months. | 12 months after starting weight management program
  All enrolled subjects will be weighed in pounds and the difference from baseline to 12 months will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bell, MD, Principal Investigator — Sanford Health
Locations (2):
- United States (2):
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Gynecological Oncology clinic, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoedjes M, van Stralen MM, Joe STA, Rookus M, van Leeuwen F, Michie S, Seidell JC, Kampman E. Toward the optimal strategy for sustained weight loss in overweight cancer survivors: a systematic review of the literature. J Cancer Surviv. 2017 Jun;11(3):360-385. doi: 10.1007/s11764-016-0594-8. Epub 2017 Jan 18. PMID 28097452
- [Background] Linkov F, Goughnour SL, Ma T, Xu Z, Edwards RP, Lokshin AE, Ramanathan RC, Hamad GG, McCloskey C, Bovbjerg DH. Changes in inflammatory endometrial cancer risk biomarkers in individuals undergoing surgical weight loss. Gynecol Oncol. 2017 Oct;147(1):133-138. doi: 10.1016/j.ygyno.2017.07.144. Epub 2017 Aug 7. PMID 28797697
- [Background] Luo J, Hendryx M, Chlebowski RT. Intentional weight loss and cancer risk. Oncotarget. 2017 Sep 6;8(47):81719-81720. doi: 10.18632/oncotarget.20671. eCollection 2017 Oct 10. No abstract available. PMID 29137210
- [Background] Massetti GM, Dietz WH, Richardson LC. Excessive Weight Gain, Obesity, and Cancer: Opportunities for Clinical Intervention. JAMA. 2017 Nov 28;318(20):1975-1976. doi: 10.1001/jama.2017.15519. No abstract available. PMID 28973170
- [Background] McCarroll ML, Armbruster S, Frasure HE, Gothard MD, Gil KM, Kavanagh MB, Waggoner S, von Gruenigen VE. Self-efficacy, quality of life, and weight loss in overweight/obese endometrial cancer survivors (SUCCEED): a randomized controlled trial. Gynecol Oncol. 2014 Feb;132(2):397-402. doi: 10.1016/j.ygyno.2013.12.023. Epub 2013 Dec 22. PMID 24369301
- [Background] McCarroll ML, Armbruster S, Pohle-Krauza RJ, Lyzen AM, Min S, Nash DW, Roulette GD, Andrews SJ, von Gruenigen VE. Feasibility of a lifestyle intervention for overweight/obese endometrial and breast cancer survivors using an interactive mobile application. Gynecol Oncol. 2015 Jun;137(3):508-15. doi: 10.1016/j.ygyno.2014.12.025. Epub 2015 Feb 11. PMID 25681782
- [Background] Steele CB, Thomas CC, Henley SJ, Massetti GM, Galuska DA, Agurs-Collins T, Puckett M, Richardson LC. Vital Signs: Trends in Incidence of Cancers Associated with Overweight and Obesity - United States, 2005-2014. MMWR Morb Mortal Wkly Rep. 2017 Oct 3;66(39):1052-1058. doi: 10.15585/mmwr.mm6639e1. PMID 28981482
- [Background] Yu J, Feng Q, Wong SH, Zhang D, Liang QY, Qin Y, Tang L, Zhao H, Stenvang J, Li Y, Wang X, Xu X, Chen N, Wu WK, Al-Aama J, Nielsen HJ, Kiilerich P, Jensen BA, Yau TO, Lan Z, Jia H, Li J, Xiao L, Lam TY, Ng SC, Cheng AS, Wong VW, Chan FK, Xu X, Yang H, Madsen L, Datz C, Tilg H, Wang J, Brunner N, Kristiansen K, Arumugam M, Sung JJ, Wang J. Metagenomic analysis of faecal microbiome as a tool towards targeted non-invasive biomarkers for colorectal cancer. Gut. 2017 Jan;66(1):70-78. doi: 10.1136/gutjnl-2015-309800. Epub 2015 Sep 25. PMID 26408641
- [Background] Zitvogel L, Ma Y, Raoult D, Kroemer G, Gajewski TF. The microbiome in cancer immunotherapy: Diagnostic tools and therapeutic strategies. Science. 2018 Mar 23;359(6382):1366-1370. doi: 10.1126/science.aar6918. PMID 29567708